CLINICAL TRIAL: NCT00858403
Title: Phase II Study of Dasatinib in Advanced Non-small Cell Lung Cancer With Ex Vivo and In Vivo Assessment of Tumor Target Modulation
Brief Title: Dasatinib in Advanced Non-small Cell Lung Cancer (NSCL) With Ex Vivo and In Vivo Assessment of Tumor Target Modulation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15656; CA180214 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2011-09-07 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Lung Cancer
Keywords: Advanced Non-small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with Dasatinib (Experimental): Dasatinib 140 mg orally (po) every day starting Day #1, continuous dosing. This dose was chosen based on the current experience in patients with solids tumors who have had prior chemotherapy.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Take tablets of Dasatinib by mouth once a day.
  Other Names: SPRYCEL®

SUMMARY:
The main purpose of this study is to learn how patients with Advanced Non-Small Cell Lung Cancer (NSCLC) respond to the study drug Dasatinib. The study drug, Dasatinib, has been approved by the U.S. Food and Drug Administration (FDA) for treatment of leukemia, but has not been approved for the treatment of other kinds of cancer. The use of Dasatinib in this study is considered experimental.

DETAILED DESCRIPTION:
Cycle 1 Day 1 (C1D1): Patients will have complete history and physical (H&P), complete blood count (CBC), complete metabolic panel (CMP) and electrocardiogram (EKG) on day 1. Each cycle is 28 days. The C1D1 EKG can be omitted if the patient has no new cardiac symptoms and has not starting taking any medication known to affect QT corrected for heart rate (QTc) prolongation. Any residual toxicity from prior therapy for cancer will be recorded. Blood will be drawn for assessment of serum markers. The patient will begin dasatinib at the starting C1D1 on a daily basis.

Cycle 1 Day 10-20 (C1D10-20): Patients will have a second biopsy to obtain additional tumor material to examine biological effects of dasatinib on signaling pathways. Dasatinib will be taken first thing in the morning and the patient will log the time. Blood will also be drawn for pharmacokinetic assessments of dasatinib levels in plasma and the time recorded. Four FNA aspirates and 2 core biopsies can be obtained either at the bedside for palpable lesions or through appropriate image-guided techniques (CT or US) at the discretion of the treating physician in consultation with radiology. The time of the biopsy will be recorded. One core biopsy should be immediately fixed in formalin and the other core biopsy should be snap frozen in liquid nitrogen.

Cycle 2 Day 1 (C2D1): Patients will be seen by the treating physician and have complete H&P, CBC, and CMP. Blood will be drawn for assessment of serum markers. Toxicity of dasatinib will be assessed. The patient will continue to take daily doses of dasatinib on a daily basis.

Cycle 2 Day 22 (C2D22): Patients will undergo reevaluation for tumor measurements. This assessment can occur on C2D22 ±7 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented diagnosis of NSCLC that is advanced/metastatic (Stage IIIB/IV).
* Performance Status (ECOG) 0-2
* Previous chemotherapy with the exception of dasatinib. Patients who have had any type of previous chemotherapy regimens for non-small cell lung cancer are eligible.
* Adequate Organ Function:

  * Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN)
  * Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN
  * Serum Na, K+, Mg2+, Phosphate and Ca2+≥ Lower Limit of Normal (LLN)
  * Serum Creatinine < 1.5 time the institutional ULN
  * Hemoglobin, Neutrophil count, Platelets, prothrombin time (PT), partial thromboplastin time (PTT) all Grade 0-1
* Ability to take oral medication
* Concomitant Medications:

  * Agree to discontinue St. Johns Wort while receiving dasatinib therapy
  * Agree that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
* Women of childbearing potential (WOCBP):

  * A negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration
  * Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped Prior to study enrollment.
* Signed written informed consent including a HIPAA form according to institutional Guidelines

Exclusion Criteria:

* No malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 years.
* Prior dasatinib therapy.
* Concurrent medical condition which may increase the risk of toxicity, including:

  * Patients with severe pulmonary disease that increases the risk of toxicity related to dasatinib-induced pleural effusions. This includes chronic obstructive pulmonary disease or pleural effusions (malignant or benign) requiring chronic oxygen therapy or patients that have had prior pneumonectomy. Patients that have a pulmonary embolism and require oxygen therapy will be excluded but not those patients who have a pulmonary embolism but do not require oxygen therapy. Patients with active pleural effusions not controlled with pleurodesis will be excluded.
* Cardiac Symptoms; any of the following should be considered for exclusion:

  * Uncontrolled angina, congestive heart failure or MI within (6 months)
  * Diagnosed congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
  * Patients with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders
  * Diagnosed acquired bleeding disorder within one year
  * Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding
* Concomitant Medications, any of the following should be considered for exclusion:

  * Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)

    1. quinidine, procainamide, disopyramide
    2. amiodarone, sotalol, ibutilide, dofetilide
    3. erythromycin, clarithromycin
    4. chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
    5. cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
* Women:

  * unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug,or
  * have a positive pregnancy test at baseline
  * pregnant or breastfeeding
* Prisoners or persons who are compulsorily detained (involuntarily incarcerated)for treatment of either a psychiatric or physical (e.g., infectious) illness
* Patients on systemic anticoagulation at risk of bleeding related to tumor biopsy that cannot be off anticoagulation per the discretion of their physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Haura, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Dasatinib
Started | 7
Completed | 2
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 7
Age, Customized [Number; unit: participants]
  Between 40 and 49 years | 1
  Between 60 and 69 years | 4
  Between 70 and 79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Progressors vs. Non-progressors With Tumor Response
Description: We planned to assess whether the extent of inhibition of extracellular signal-regulated protein kinase (ERK) phosphorylation in lung cancer cells exposed ex vivo to dasatinib significantly differed between patients categorized as progressors or non-progressors through standard Response Evaluation Criteria In Solid Tumors (RECIST)
Time Frame: 1 year, 4 months
Population: The low accrual of 7 participants prevented us from completing the planned analysis. Target accrual was 40.
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Response to Dasatinib
Description: We planned to estimate the single agent response rate to dasatinib in this patient population
Time Frame: 1 year, 4 months
Population: The low accrual of 7 participants prevented us from completing the planned analysis. Target accrual was 40.
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) at 6 Months
Description: We planned to estimate the 6 month progression free survival rate of dasatinib in this patient population.
Time Frame: 1 year, 4 months
Population: We were able to assess 4 of the 7 participants at 6 months.
Measure: Number; unit: Participants
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 4
Participants | 1

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: We evaluated toxicity of dasatinib in this patient population.
Time Frame: 1 year, 4 months
Measure: Number; unit: Participants
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 7
Participants | 3

5. Secondary Outcome: Number of Participant Progressors vs. Non-Progressors With Inhibition Response
Description: We planned to assess whether the extent of inhibition of proto-oncogene tyrosine-protein kinase (SRC) and protein kinase B (Akt) phosphorylation in lung cancer cells exposed ex vivo and in vivo to dasatinib significantly differs between patients categorized as progressors or non-progressors through standard RECIST criteria.
Time Frame: 1 year, 4 months
Population: The low accrual of 7 participants prevented us from completing the planned analysis. Target accrual was 40.
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation Between Extent of Inhibition and Concentration of Dasatinib
Description: We planned to explore whether the extent of inhibition of ERK, SRC and Akt phosphorylation in lung cancer cells exposed ex vivo to dasatinib will correlate with the drug concentration of dasatinib.
Time Frame: 1 year, 4 months
Population: The low accrual of 7 participants prevented us from completing the planned analysis. Target accrual was 40.
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Correlation Between Mutation and Inhibition and to Disease Control Rate and Response
Description: To analyze Kras and epidermal growth factor receptor (EGFR) mutation and their correlation to the ERK pathway inhibition and to disease control rate and response.
Time Frame: 1 year, 4 months
Population: The low accrual of 7 participants prevented us from completing the planned analysis. Target accrual was 40.
Arm/Group | Treatment With Dasatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Description: From first participant on study date to last participant off study date.
Arm/Group | Treatment With Dasatinib
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Dasatinib (N=7)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) — Grade 3 - unlikely to be related
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) — Grade 4 - unrelated
Death Due to Disease Progression (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5 - unlikely to be related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 4 - unrelated
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3 - unrelated
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3 - probably related
Fatigue (General disorders) | 1 (1) — Grade 3 - probably related
Fever in absence of neutropenia (General disorders) | 1 (1) — Grade 2 - unrelated
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 4 - unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment With Dasatinib (N=7)
Abdomen Pain (General disorders) | 1 (1) — Grade 1 - unlikely to be related
Anorexia (Metabolism and nutrition disorders) | 1 (1) — Grade 1 - possibly related
Anorexia (Metabolism and nutrition disorders) | 1 (1) — Grade 2 - possibly related
Back Pain (General disorders) | 1 (1) — Grade 1 - unrelated
Blurred Vision (Eye disorders) | 1 (1) — Grade 1 - possibly related
Constipation (Gastrointestinal disorders) | 1 (1) — Grade 1 - possibly related
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1 - possibly related
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1 - unrelated
Creatinine (Renal and urinary disorders) | 1 (1) — Grade 1 - unlikely to be related
Dehydration (Gastrointestinal disorders) | 1 (1) — Grade 3 - unrelated
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 1 - possibly related
Dizziness (General disorders) | 1 (1) — Grade 1 - possibly related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1 - related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3 - related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1 - probably related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 2 - related
Dyspnea - With Exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 2 - unrelated
Dysuria (Renal and urinary disorders) | 1 (1) — Grade 2 - possibly related
Edema - Limb (Blood and lymphatic system disorders) | 1 (1) — Grade 1 - possibly related
Fatigue (General disorders) | 1 (1) — Grade 2 - probably related
Fatigue (General disorders) | 1/1 (1) — Grade 1 - probably related
Fever (General disorders) | 1 (1) — Grade 1 - unlikely to be related
Headaches (General disorders) | 1 (1) — Grade 1 - possibly related
Hemoglobin - Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 2 - probably related
Hemorrhage - Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1 - unrelated
Insomnia (General disorders) | 1 (1) — Grade 2 - unrelated
Nausea - Intermittent (General disorders) | 1 (1) — Grade 1 - probably related
Nausea - Intermittent (Gastrointestinal disorders) | 1 (1) — Grade 2 - possibly related
Pleural Effusion - Intermittent (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 2 - related
Voice Hoarseness (General disorders) | 1 (1) — Grade 1 - unlikely to be related
Vomiting - Intermittent (Gastrointestinal disorders) | 1 (1) — Grade 2 - possibly related

LIMITATIONS AND CAVEATS:
The low accrual of 7 participants prevented us from completing the planned analysis. Target accrual was 40.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes